CLINICAL TRIAL: NCT05133011
Title: Efficacy of Force Sensing Resistor Assisted Physical Therapy Program for Obstructive Sleep Apnea With Low-responsiveness of Oropharyngeal Muscle Patients After Tongue Base Reduction Surgery：Establishment of Precision Medicine
Brief Title: Force Sensing Resistor for Obstructive Sleep Apnea Patients After Tongue Base Reduction Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cheng-Kung University Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-BR-109-058
Record Dates: First submitted 2021-11-14; First posted 2021-11-24 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2021-11

CONDITIONS: Sleep Apnea, Obstructive
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low muscle strength (Experimental): The participants underwent before tongue base reduction surgery used Iowa Oral Performance Instrument (IOPI) system test upper tongue muscle strength were the last 5%
  Interventions: Procedure: Tongue base reduction surgery
- Normal groups (Experimental): The participants underwent before tongue base reduction surgery used Iowa Oral Performance Instrument (IOPI) system test upper tongue muscle strength were greater than 5%
  Interventions: Procedure: Tongue base reduction surgery

INTERVENTIONS:
Procedure: Tongue base reduction surgery — Tongue base reduction surgery which remove the extra soft tissue of the base of the tongue and soft palate in this study

SUMMARY:
Obstructive sleep apnea syndrome (OSA) is a sleep-related breathing disorder defined by repetitive episodes of apnea and hypopnea. These traits include anatomical (narrow/crowded/collapsible upper airway) and nonanatomical (waking up too easily during airway narrowing [a low respiratory arousal threshold], ineffective or reduced pharyngeal dilator muscle activity during sleep, and unstable ventilatory control [high loop gain]) components. Oropharyngeal training reduces the snoring times, Apnea-hypopnea Index (AHI) and daytime sleepiness. There is lack of good evaluating tools to distinguish different phenotypes of OSA and the efficacy of combined therapy. The purposes of our study are (1) to evaluate OSA patient by using Polysomonogrphy (PSG), force sensing resistor (FRS), Drug induce sleep endoscopy (DISE) and CT and muscle strength testing, (2) to know the exercise times by using FSR and (3) the efficacy of exercise in different groups.

DETAILED DESCRIPTION:
Subjects who are newly diagnosed with mild to severe OSA (AHI >5/h), and the physician will explain the treatment programs to every subject. By the result of muscle strength testing, the subjects will be classified as low muscle strength and normal groups. The myofunctional therapy program will begin at 6 week after surgery, and subjects will undergo 12 weeks of the home-based oropharyngeal myofunctional therapeutic training. During the training intervention period, subjects will be interviewed one time per week for adjusting the treatment intensity.

Expected results：The hypothesis of this study is the efficacy of exercise would be less in the low muscle strength OSA patient than normal.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of mild to severe OSA in the past year
* Agree to receive Transoral Robotic Surgery (TORS)
* Age between 20-65 years old.

Exclusion Criteria:

* Body Mass Index ≧ 32
* Drug abuse within one year
* Pregnant
* Severe obstructive or restrictive lung disease
* A history of malignancy or infection of the head and neck region and laryngeal trauma
* Craniofacial malformation
* Stroke
* Neuromuscular disease
* Heart failure
* Coronary artery disease
* Ongoing or uncontrolled chronic diseases
* Combine central or mixed types sleep apnea syndrome
* Other non-breath related sleep disorder.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-22 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Apnea and Hypopnea index (AHI) at post op 6 weeks and 18 weeks | through study completion, an average of 18 weeks
  Polysomnography included electroencephalographic, electro-oculographic, thoracic and abdominal respiratory inductance plethysmography and body position sensor to confirm the sleeping stage in one-night observation. Above measurements will be aggregated to arrive AHI.
Change from Baseline Volume from hard palate to the base of epiglottis in computer tomography (CT) at post op 6 weeks and 18 weeks | through study completion, an average of 18 weeks
  All patients underwent CT in a supine position. Each patient was instructed to maintain his/her tongue in the resting position, without swallowing, during CT. Volume from hard palate to the base of epiglottis was measured.
Change from Baseline Cross section area on the tip of epiglottis in computer tomography (CT) at post op 6 weeks and 18 weeks | through study completion, an average of 18 weeks
  All patients underwent CT in a supine position. Each patient was instructed to maintain his/her tongue in the resting position, without swallowing, during CT. Cross section area on the tip of epiglottis was measured.
Change from Baseline Anterior to posterior distance on the tip of epiglottis in computer tomography (CT) at post op 6 weeks and 18 weeks | through study completion, an average of 18 weeks
  All patients underwent CT in a supine position. Each patient was instructed to maintain his/her tongue in the resting position, without swallowing, during CT. Anterior to posterior distance on the tip of epiglottis was measured.
Change from Baseline Lateral distance on the tip of epiglottis in computer tomography (CT) at post op 6 weeks and 18 weeks | through study completion, an average of 18 weeks
  All patients underwent CT in a supine position. Each patient was instructed to maintain his/her tongue in the resting position, without swallowing, during CT. Anterior to posterior distance on the tip of epiglottis was measured.
Change from Baseline Drug-induced sleep endoscopy (DISE) at post op 6 weeks and 18 weeks | through study completion, an average of 18 weeks
  DISE was carried out by an experienced ENT surgeon in a semi-dark and quiet operating room with the patient supine lying on a hospital bed. Artificial sleep was induced by intravenous injection of propofol and midazolam (bolus injection of 1.5 mg) through a target-controlled infusion system (1.5 to 3.0 lg/mL), intending to the transition to unconsciousness with beginning of snoring and with the examiner evaluating decreased muscle reflexes of the eyelid. The severity of collapse in the upper airway was assessed by the surgeon.
Change from Baseline Muscle Strength of Jaw at post op 6 weeks and 18 weeks | through study completion, an average of 18 weeks
  Muscle strength of jaw was measured with a 'handheld' dynamometer (MicroFET○R2, Hoggan Scientific, USA) mounted on an adapted ophthalmic examination frame, to avoid alterations in chin and head position and to ensure consistent compression.
Change from Baseline Muscle strength of tongue at post op 6 weeks and 18 weeks | through study completion, an average of 18 weeks
  The muscle strength of the tongue was evaluated by the IOPI system, model 2.2 (Northwest, Co., LLC, Carnation, WA, USA).

CONTACTS AND LOCATIONS:
Overall Officials: Ching-Hsia Hung, PhD, Principal Investigator — Department of physical therapy, National Cheng Kung University
Locations (1):
- National Cheng Kung University Hospital, Tainan, Please Select, Taiwan